CLINICAL TRIAL: NCT01420757
Title: Laparoscopic Versus Open Incisional Hernia Repair : A Randomized Clinical Trial
Brief Title: Laparoscopic Versus Open Incisional Hernia Repair
Acronym: COLIBRI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, hasan eker, Prof. Dr. J.F. Lange, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COLIBRI trial
Record Dates: First submitted 2011-08-18; First posted 2011-08-22 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Postoperative Pain; Complications; Recurrence
Keywords: operation time; length of hospital stay
MeSH Terms: conditions — Pain, Postoperative; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- open (Active Comparator): open incisional hernia repair
  Interventions: Procedure: incisional hernia repair
- laparoscopic (Active Comparator): laparoscopic incisional hernia repair
  Interventions: Procedure: incisional hernia repair

INTERVENTIONS:
Procedure: incisional hernia repair — Tension-free open or laparoscopic incisional hernia repair

SUMMARY:
Primary closure of incisional hernia without the use of a mesh shows recurrence rates of up to 54%. If a mesh is used, the defect can be closed tension-free. Using this method, recurrence rates have been reduced to 8-21%. Laparoscopic correction of incisional hernia is a relatively new technique in which the mesh is positioned intraperitoneally. Research has shown that this procedure is technical feasible and may have benefits for the patients.

The ongoing debate about the merits of endoscopic versus open incisional hernia repair prompts the need for a level 1 randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* hernia diameter between 3 and 15 cm
* location at the ventral abdominal wall at least 5cm from costae and inguinal area
* indication for elective repair
* age of 18 years or older
* written informed consent.

Exclusion Criteria:

* contraindication for pneumoperitoneum
* an absolute contraindication for general anesthesia
* history of open abdomen treatment
* patients participating in other trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 1999-05; Primary Completion 2006-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 4 weeks

SECONDARY OUTCOMES:
Postoperative analgesics use | 1 week
complications | 4 weeks
operation time | 1 day
length of hospital stay | 4 weeks
recurrence | 5 years
mortality | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: J.F. Lange, MD, PhD, Principal Investigator — Erasmus Medical Center